CLINICAL TRIAL: NCT03993535
Title: Clinical, Neurocognitive and Neuroimaging Variables Associated With Response to Treatment in Patients With OCD
Brief Title: Predicting Treatment Response in Patients With OCD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: University of Stellenbosch (Other); Columbia University (Other); National Institute of Mental Health and Neuro Sciences, India (Other); Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Roseli Gedanke Shavitt, Director, Obsessive-Compulsive Spectrum Disorders Program, Institute of Psychiatry, Hospital of Clinics, University of Sao Paulo School of Medicine, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 68743617800000068
Record Dates: First submitted 2019-06-13; First posted 2019-06-20 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: obsessive-compulsive disorder; predictors; neuroimaging
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Intervention Model Description: 12-month naturalistic follow-up of open treatment with evidence-based pharmacologic agents (SSRIs) or cognitive-behavioral therapy (CBT) for OCD
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- SSRI or cognitive behavioral therapy (Other): selective serotonin reuptake inhibitors (fluoxetine, sertraline, citalopram, escitalopram, paroxetine or fluvoxamine) or cognitive-behavioral therapy, depending on availability and patient preference
  Interventions: Drug: selective serotonin reuptake inhibitor

INTERVENTIONS:
Drug: selective serotonin reuptake inhibitor — open treatment based on patient preference and treatment availability
  Other Names: CBT

SUMMARY:
This study consists of a naturalistic follow-up of subjects with Obsessive-Compulsive Disorder (OCD) that have participated in a global study investigating brain signatures of OCD funded by the National Institutes of Mental Health (RO1MH113250), with the following participant sites: the US (Columbia University, PI: Helen Blair Simpson), Brazil (University of Sao Paulo, PIs: Euripedes Miguel and Roseli G Shavitt), India (National Institutes of Mental Health, PI: Janardhan Reddy), The Netherlands (VU Amsterdam Medical Center, PI: Odile van den Heuvel), and South Africa (University of Cape Town, PI: Dan Stein; Stellenbosch University, PI: Christine Lochner). In this cross-sectional study, two-hundred and fifty unmedicated subjects with OCD (50 per site) will be assessed for clinical, neurocognitive and neuroimaging data. After completion of this study, participants willing to receive evidence-based treatments for OCD will be treated with the available resources in each site and will be assessed for treatment response status periodically, with a final assessment after 1 year of naturalistic follow-up. At this point, we will investigate baseline clinical, neurocognitive and neuroimaging variables associated with the treatment response status.

DETAILED DESCRIPTION:
This study aims to investigate clinical, neurocognitive and neuroimaging variables associated with response to conventional treatments in adults with OCD.

Study design:

* 0-52 weeks: open-label trial of a selective serotonin reuptake inhibitor (SSRI) (preferably sertraline - easily available in the public network, usually well tolerated) up to the maximum recommended or tolerated dose (e.g., titration: start with 50mg/day, then add 50mg/day per week up to 200mg/day, if sertraline); patients who prefer to be treated with cognitive-behavioral therapy (CBT) will be given this option whenever CBT is available.
* treatment will be delivered under naturalistic conditions, tailored according to the needs, preference, and availability. Subjects will be called up for follow-up assessments at 3, 6, 9 and 12 months after baseline assessments. The instruments to be used at follow-up are the YBOCS and CGI scales.
* Response criteria: the definitions of a recent international expert consensus will be adopted (Mataix-Cols. et al., 2016). A positive response will be considered as at least 35% reduction in baseline Yale-Brown Obsessive-Compulsive Scale (YBOCS) scores plus a Clinical Global Impression-Improvement (CGI-I) rating of 1 ("very much improved") or 2 ("much improved"), lasting for at least one week. We will also rate the CGI - severity. Partial response will correspond to a greater than 25% but less than 35% reduction in Y-BOCS scores plus a CGI-I rating of at least 3 ("minimally improved"), lasting for at least one week.

Subjects:

• All participants assessed for clinical, neurocognitive and neuroimaging data in the global brain signatures study who are willing to receive evidence-based treatment for OCD.

Assessments:

* Baseline: clinical, neurocognitive and neuroimaging protocols.

  1. Clinical: interviewer-delivered and self-report measures to determine: socio-demographic data, past medical history, psychiatric family history, psychiatric diagnoses, OCD symptom dimensions, the severity of OCD, insight into OCD, sensory phenomena, the severity of depression and anxiety symptoms, severity of compulsive-impulsive behaviors, level of disability
  2. Neurocognitive: executive function, emotional regulation, memory
  3. Neuroimaging: structural MRI, resting-state functional MRI (rs-fMRI), Diffusion Tensor Imaging (DTI)
* Months 3, 6, 9 and 12: YBOCS checklist and past week severity; CGI - improvement subscale, relative to baseline; CGI - severity subscale; assessments can be in person or by phone, by the same independent evaluator at the different time points
* 1 year: treatment history form, YBOCS severity and checklist, Impulsive-Compulsive Behaviors Checklist (ICBC), Obsessive-Compulsive Inventory-Revised (OCI-R), Hamilton Depression Scale (HAM-D), Hamilton Anxiety Scale (HAM-A), World Health Organization Disability Assessment Schedule (WHODAS), CGI.

Hypotheses (built from the literature): the following variables (as assessed at baseline) will show an association with response to treatment:

Clinical:

1. duration of untreated illness (Alarcon et al., 1993; Ravizza et al., 1995; Stein et al., 2001);
2. comorbidity: presence of comorbid social anxiety disorder (Carrasco et al., 1992), depressive disorders (Jakubovski et al., 2013); Post-Traumatic Stress Disorder (PTSD) (Shavitt et al., 2010);
3. level of insight (Erzegovesi et al., 2001);
4. symptom dimension: presence and severity of symmetry, contamination and hoarding dimensions (Alarcon et al., 1993; Ferrão et al., 2006; Mataix-Cols et al., 1999; Hazari et al., 2016)

Neurocognitive: decision making, verbal IQ (D'Alcante et al., 2012), verbal memory/learning (D'Alcante et al., 2012), inhibitory control and mental flexibility tasks (Flessner et al., 2010; Hazari et al., 2016).

Neuroimaging:

I. Structural: brain volumes in the orbitofrontal cortex, anterior cingulate, striatum, dorsolateral and dorsomedial prefrontal cortex (Yun et al., 2015), insula (Yun et al., 2015), thalamus, hippocampus, pituitary gland (Atmaca et al., 2016), amygdala (Szeszko et al., 2004), and cerebellum.

II. Structural connectivity (Diffusion Tensor Imaging - DTI): fractional anisotropy measures in the corpus callosum, the internal capsule, white matter in the area superolateral to the right caudate, bilateral cingulum, superior longitudinal fasciculus, and inferior longitudinal fasciculus (Cannistraro et al., 2007; Szeszko wt al., 2005; Yoo et al., 2007; Garibotto et al., 2010).

III. Functional connectivity (rs-fMRI): patterns of activation and connectivity in frontal-striatal (central executive), parietal, occipital, cerebellar, and insula-limbic (saliency) networks (Shin et al., 2014; Bhikram et al., 2016; Nakao et al., 2005; Sanematsu et al., 2010) IV. Exploratory: multimodal analyses of prediction

Analyses plan: parametric and non-parametric tests will be employed as indicated.

ELIGIBILITY:
Inclusion Criteria:

* Principal DSM-5 diagnosis of OCD
* Y-BOCS ≥ 16
* No psychotropic meds for the last 6 weeks, with the exception of PRN sleeping meds (e.g., zolpidem or trazodone up to 50 mg) and benzos, as long as not within the past week or during study participation
* No CBT/EXRP focused on OCD within the past 6 weeks
* Capable of providing informed consent

Exclusion Criteria:

* Lifetime diagnosis of psychotic disorder, bipolar disorder, anorexia nervosa, autism spectrum disorder with IQ < 80, Tourette Disorder
* Current chronic tic disorder (current = in the past 12 months)
* Current substance-related and addictive disorders, including nicotine (current = in the past 12 months)
* Current binge-eating disorder or bulimia (current = in the past 12 months)
* Acute risk of suicide
* Female who is pregnant
* Major medical or neurological problems (including head injury with loss of consciousness) Presence of metallic devices or dental braces
* IQ < 80
* Cigarette use: more than 5 per day
* Alcohol use: more than 2 drinks per day for women and more than 3 drinks per day for men, Marijuana use: more than once per week

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
response status | 12 months
  severity of OCD as measured by the Yale-Brown Obsessive-Compulsive Scale. The final score of this scale is a sum of 10 items, ranging from 0 to 40. The higher the score, the more severe the clinical picture. The ten items refer to ten questions, five regarding obsessions and five regarding compulsions. The questions assess time, distress, interference, resistance and control over the symptoms. Each question can be rated from 0 (= none) to 4 (most severe).
level of improvement | 12 months
  measured by the Clinical Global Impression Scale - severity and improvement subscales. The severity subscale can be rated from 1 to 7, a higher score corresponding to more severe symptoms. The improvement subscale can also be rated from 1 to 7, a greater score corresponding to lesser improvement. Scores are given individually to each subscale, in absolute numbers (1 to 7)

CONTACTS AND LOCATIONS:
Overall Officials: Roseli G Shavitt, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (4):
- Center for OCD and Related Disorders, New York State Psychiatric Institute/Columbia University Medical Center, New York, New York, United States
- Institute of Psychiatry - Hospital of Clinics - University of São Paulo, São Paulo, Brazil
- OCD Clinic, Department of Psychiatry, National Institute of Mental Health and Neurosciences (NIMHANS), Bangalore, India
- Faculty of Medicine and Health Sciences, Department of Psychiatry, Stellenbosch University, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alarcon RD, Libb JW, Spitler D. A predictive study of obsessive-compulsive disorder response to clomipramine. J Clin Psychopharmacol. 1993 Jun;13(3):210-3. PMID 8354737
- [Background] Atmaca M, Mermi O, Yildirim H, Gurok MG. Orbito-frontal cortex and thalamus volumes in obsessive-compulsive disorder before and after pharmacotherapy. Brain Imaging Behav. 2016 Sep;10(3):669-74. doi: 10.1007/s11682-015-9426-0. PMID 26311393
- [Background] Baer L, Jenike MA, Black DW, Treece C, Rosenfeld R, Greist J. Effect of axis II diagnoses on treatment outcome with clomipramine in 55 patients with obsessive-compulsive disorder. Arch Gen Psychiatry. 1992 Nov;49(11):862-6. doi: 10.1001/archpsyc.1992.01820110026003. PMID 1444723
- [Background] Bhikram TP, Farb NA, Ravindran LN, Papadopoulos YG, Conn DK, Pollock BG, Ravindran AV. The Effect of Intravenous Citalopram on the Neural Substrates of Obsessive-Compulsive Disorder. J Neuropsychiatry Clin Neurosci. 2016 Summer;28(3):243-7. doi: 10.1176/appi.neuropsych.15090213. Epub 2016 Mar 28. PMID 27019066
- [Background] Cannistraro PA, Makris N, Howard JD, Wedig MM, Hodge SM, Wilhelm S, Kennedy DN, Rauch SL. A diffusion tensor imaging study of white matter in obsessive-compulsive disorder. Depress Anxiety. 2007;24(6):440-6. doi: 10.1002/da.20246. PMID 17096398
- [Background] Carrasco JL, Hollander E, Schneier FR, Liebowitz MR. Treatment outcome of obsessive compulsive disorder with comorbid social phobia. J Clin Psychiatry. 1992 Nov;53(11):387-91. PMID 1459968
- [Background] D'Alcante CC, Diniz JB, Fossaluza V, Batistuzzo MC, Lopes AC, Shavitt RG, Deckersbach T, Malloy-Diniz L, Miguel EC, Hoexter MQ. Neuropsychological predictors of response to randomized treatment in obsessive-compulsive disorder. Prog Neuropsychopharmacol Biol Psychiatry. 2012 Dec 3;39(2):310-7. doi: 10.1016/j.pnpbp.2012.07.002. Epub 2012 Jul 10. PMID 22789662
- [Background] Erzegovesi S, Cavallini MC, Cavedini P, Diaferia G, Locatelli M, Bellodi L. Clinical predictors of drug response in obsessive-compulsive disorder. J Clin Psychopharmacol. 2001 Oct;21(5):488-92. doi: 10.1097/00004714-200110000-00006. PMID 11593074
- [Background] Flessner CA, Allgair A, Garcia A, Freeman J, Sapyta J, Franklin ME, Foa E, March J. The impact of neuropsychological functioning on treatment outcome in pediatric obsessive-compulsive disorder. Depress Anxiety. 2010 Apr;27(4):365-71. doi: 10.1002/da.20626. PMID 19842168
- [Background] Garibotto V, Scifo P, Gorini A, Alonso CR, Brambati S, Bellodi L, Perani D. Disorganization of anatomical connectivity in obsessive compulsive disorder: a multi-parameter diffusion tensor imaging study in a subpopulation of patients. Neurobiol Dis. 2010 Feb;37(2):468-76. doi: 10.1016/j.nbd.2009.11.003. Epub 2009 Nov 11. PMID 19913616
- [Background] Hazari N, Narayanaswamy JC, Arumugham SS. Predictors of response to serotonin reuptake inhibitors in obsessive-compulsive disorder. Expert Rev Neurother. 2016 Oct;16(10):1175-91. doi: 10.1080/14737175.2016.1199960. Epub 2016 Jun 30. PMID 27282021
- [Background] Jakubovski E, Diniz JB, Valerio C, Fossaluza V, Belotto-Silva C, Gorenstein C, Miguel E, Shavitt RG. Clinical predictors of long-term outcome in obsessive-compulsive disorder. Depress Anxiety. 2013 Aug;30(8):763-72. doi: 10.1002/da.22013. Epub 2012 Oct 25. PMID 23109056
- [Background] Jenike MA, Baer L, Minichiello WE, Schwartz CE, Carey RJ Jr. Concomitant obsessive-compulsive disorder and schizotypal personality disorder. Am J Psychiatry. 1986 Apr;143(4):530-2. doi: 10.1176/ajp.143.4.530. PMID 3953896
- [Background] Mataix-Cols D, Rauch SL, Manzo PA, Jenike MA, Baer L. Use of factor-analyzed symptom dimensions to predict outcome with serotonin reuptake inhibitors and placebo in the treatment of obsessive-compulsive disorder. Am J Psychiatry. 1999 Sep;156(9):1409-16. doi: 10.1176/ajp.156.9.1409. PMID 10484953
- [Background] Mataix-Cols D, Fernandez de la Cruz L, Nordsletten AE, Lenhard F, Isomura K, Simpson HB. Towards an international expert consensus for defining treatment response, remission, recovery and relapse in obsessive-compulsive disorder. World Psychiatry. 2016 Feb;15(1):80-1. doi: 10.1002/wps.20299. No abstract available. PMID 26833615
- [Background] Nakao T, Nakagawa A, Yoshiura T, Nakatani E, Nabeyama M, Yoshizato C, Kudoh A, Tada K, Yoshioka K, Kawamoto M, Togao O, Kanba S. Brain activation of patients with obsessive-compulsive disorder during neuropsychological and symptom provocation tasks before and after symptom improvement: a functional magnetic resonance imaging study. Biol Psychiatry. 2005 Apr 15;57(8):901-10. doi: 10.1016/j.biopsych.2004.12.039. PMID 15820711
- [Background] Ravizza L, Barzega G, Bellino S, Bogetto F, Maina G. Predictors of drug treatment response in obsessive-compulsive disorder. J Clin Psychiatry. 1995 Aug;56(8):368-73. PMID 7635854
- [Background] Sanematsu H, Nakao T, Yoshiura T, Nabeyama M, Togao O, Tomita M, Masuda Y, Nakatani E, Nakagawa A, Kanba S. Predictors of treatment response to fluvoxamine in obsessive-compulsive disorder: an fMRI study. J Psychiatr Res. 2010 Mar;44(4):193-200. doi: 10.1016/j.jpsychires.2009.08.007. Epub 2009 Sep 15. PMID 19758599
- [Background] Shavitt RG, Valerio C, Fossaluza V, da Silva EM, Cordeiro Q, Diniz JB, Belotto-Silva C, Cordioli AV, Mari J, Miguel EC. The impact of trauma and post-traumatic stress disorder on the treatment response of patients with obsessive-compulsive disorder. Eur Arch Psychiatry Clin Neurosci. 2010 Mar;260(2):91-9. doi: 10.1007/s00406-009-0015-3. PMID 20077119
- [Background] Shin NY, Lee TY, Kim E, Kwon JS. Cognitive functioning in obsessive-compulsive disorder: a meta-analysis. Psychol Med. 2014 Apr;44(6):1121-30. doi: 10.1017/S0033291713001803. Epub 2013 Jul 19. PMID 23866289
- [Background] Stein DJ, Montgomery SA, Kasper S, Tanghoj P. Predictors of response to pharmacotherapy with citalopram in obsessive-compulsive disorder. Int Clin Psychopharmacol. 2001 Nov;16(6):357-61. doi: 10.1097/00004850-200111000-00007. PMID 11712625
- [Background] Szeszko PR, MacMillan S, McMeniman M, Lorch E, Madden R, Ivey J, Banerjee SP, Moore GJ, Rosenberg DR. Amygdala volume reductions in pediatric patients with obsessive-compulsive disorder treated with paroxetine: preliminary findings. Neuropsychopharmacology. 2004 Apr;29(4):826-32. doi: 10.1038/sj.npp.1300399. PMID 14970831
- [Background] Szeszko PR, Ardekani BA, Ashtari M, Malhotra AK, Robinson DG, Bilder RM, Lim KO. White matter abnormalities in obsessive-compulsive disorder: a diffusion tensor imaging study. Arch Gen Psychiatry. 2005 Jul;62(7):782-90. doi: 10.1001/archpsyc.62.7.782. PMID 15997020
- [Background] Yoo SY, Jang JH, Shin YW, Kim DJ, Park HJ, Moon WJ, Chung EC, Lee JM, Kim IY, Kim SI, Kwon JS. White matter abnormalities in drug-naive patients with obsessive-compulsive disorder: a diffusion tensor study before and after citalopram treatment. Acta Psychiatr Scand. 2007 Sep;116(3):211-9. doi: 10.1111/j.1600-0447.2007.01046.x. PMID 17655563
- [Background] Yun JY, Jang JH, Kim SN, Jung WH, Kwon JS. Neural Correlates of Response to Pharmacotherapy in Obsessive-Compulsive Disorder: Individualized Cortical Morphology-Based Structural Covariance. Prog Neuropsychopharmacol Biol Psychiatry. 2015 Dec 3;63:126-33. doi: 10.1016/j.pnpbp.2015.06.009. Epub 2015 Jun 24. PMID 26116795